CLINICAL TRIAL: NCT05516290
Title: An In Depth Study Investigating Patterns of Patients In Congestive Heart Failure Clinical Trials
Brief Title: Evaluating Clinical Trial Experiences of Individuals With Congestive Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 85707278
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trial participation has always been substantially skewed toward certain demographic groups. However, there has been little study on whether trial qualities impact participation in either a positive or negative way. The goal of this research is to identify the characteristics that consistently restrict patients' ability to participate in or complete a trial in which they were initially interested. This data will be evaluated via a number of demographic lenses in order to find trends that could benefit future Congestive Heart Failure sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the United States
* Is 18+ years old
* Participant has a diagnosis of congestive heart failure
* Participant has enrolled in an interventional clinical for congestive heart failure (self-reported)

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form
* No diagnosis of congestive heart failure confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Congestive Heart Failure patients who are actively considering enrolling in an interventional clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patient decides to enroll in a congestive heart failure clinical trial | 3 months
Rate of patients who remain in a congestive heart failure clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

REFERENCES:
- [Background] Betkowski AS, Hauptman PJ. Update on recent clinical trials in congestive heart failure. Curr Opin Cardiol. 2000 Jul;15(4):293-303. doi: 10.1097/00001573-200007000-00015. PMID 11139094
- [Background] White M, Rouleau JL. Overview of clinical trials in congestive heart failure. Can J Cardiol. 1993 Sep;9(7):629-34. PMID 8221362
- [Background] Samman Tahhan A, Vaduganathan M, Kelkar A, Georgiopoulou VV, Kalogeropoulos AP, Greene SJ, Fonarow GC, Gheorghiade M, Butler J. Trends in Heart Failure Clinical Trials From 2001-2012. J Card Fail. 2016 Mar;22(3):171-9. doi: 10.1016/j.cardfail.2015.06.014. Epub 2015 Jun 21. PMID 26106806

DOCUMENTS (1):
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT05516290/ICF_000.pdf